CLINICAL TRIAL: NCT05362526
Title: Prevention of Pulmonary Complications Using High Flow With Tracheostomy Interface vs Conventional Oxygen Therapy in Patients After Major Head and Neck Surgery: Randomized Clinical Trial
Brief Title: High Flow vs Conventional Oxygen in Head and Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202102700; AGR00023048 (Other: UFIRST)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Disease
Keywords: Head neck surgery; heated humidification; cool humidification
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High flow with tracheostomy interface (Experimental): Patient will be placed on heated humidified high flow after surgery.
  Interventions: Device: High flow humidification
- Conventional Oxygen Therapy (Active Comparator): Pt will be placed on conventional oxygen therapy after surgery.
  Interventions: Device: Conventional cool mist aerosol humidification

INTERVENTIONS:
Device: High flow humidification — High flow is for the treatment of spontaneously breathing patients who would benefit from receiving high flow warmed and humidified respiratory gases. The subjects in this group will receive HFOT at a flow rate of 60-30 liters per minute, maximum concentration of 40%, which will be titrated by bedside nurse to maintain an oxygen saturation of 92% or greater (unless there is a history of COPD and then the clinician can recommend >88%)
  Arms: High flow with tracheostomy interface
Device: Conventional cool mist aerosol humidification — Subjects will be placed on aerosolized trach mask with cool humidification, and titrated to keep oxygen saturation >92% (unless there is a history of COPD and then the clinician can recommend >88%)
  Arms: Conventional Oxygen Therapy

SUMMARY:
Patients undergoing major head and neck surgery are at risk for postoperative pulmonary complications. The goal of this randomized clinical trial is to evaluate the effectiveness of high flow heated humidified oxygen at preventing postoperative pulmonary complications after major head and neck surgery, when compared to conventional oxygen therapy (aerosol cool mist).

DETAILED DESCRIPTION:
Participants enrolled in this study are randomly assigned to receive either conventional oxygen therapy (aerosol cool mist) or heated humidified high flow oxygen via the trach after head and neck surgery. The study team then collects information regarding clinical outcomes to explore if there are differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major head and neck surgery that includes any neck dissection
* Major head and neck surgery is defined as having a mean length of stay of three or more days, based on the diagnosis [14]
* Surgery requires an elective tracheostomy for airway protection or laryngectomy tube in the case of total laryngectomy

Exclusion Criteria:

* <18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Fernandes, MD, DMD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 consented and randomized.
Groups:
- High Flow With Tracheostomy Interface: Patient will be placed on heated humidified high flow after surgery.
  High flow humidification: High flow is for the treatment of spontaneously breathing patients who would benefit from receiving high flow warmed and humidified respiratory gases. The subjects in this group will receive HFOT at a flow rate of 60-30 liters per minute, maximum concentration of 40%, which will be titrated by bedside nurse to maintain an oxygen saturation of 92% or greater (unless there is a history of chronic obstructive pulmonary disease) and then the clinician can recommend >88%)
Period: Overall Study
Arm/Group | High Flow With Tracheostomy Interface | Conventional Oxygen Therapy
Started | 26 | 30
Completed | 24 | 25
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- HFOT (High Flow With Tracheostomy Interface): Patient will be placed on heated humidified high flow after surgery.
  High flow humidification: High flow is for the treatment of spontaneously breathing patients who would benefit from receiving high flow warmed and humidified respiratory gases. The subjects in this group will receive HFOT at a flow rate of 60-30L liters per minute, maximum concentration of 40%, which will be titrated by bedside nurse to maintain an oxygen saturation of 92% or greater (unless there is a history of COPD and then the clinician can recommend >88%)
- COT (Conventional Oxygen Therapy): Pt will be placed on conventional oxygen therapy after surgery.
  Conventional cool mist aerosol humidification: Subjects will be placed on aerosolized trach mask with cool humidification, and titrated to keep oxygen saturation >92% (unless there is a history of COPD and then the clinician can recommend >88%)
- Total: Total of all reporting groups
Arm/Group | HFOT (High Flow With Tracheostomy Interface) | COT (Conventional Oxygen Therapy) | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 5 | 15 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (13.5) | 66.8 (9.2) | 61.57 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 13 | 18 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49
Body mass index [Mean (Standard Deviation); unit: kilograms per square meter] | 26.7 (8.9) | 26.2 (6.8) | 26.469 (7.83)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Post-operative Pulmonary Complication
Description: Postoperative pulmonary complication will be defined as:
  * Atelectasis or infiltrate diagnosed by radiologist on any postoperative chest radiograph within first 14 days or discharge (whichever occurs first)
  * Pneumonia Diagnosis is suggested by a history of cough, dyspnea, pleuritic pain, or acute functional or cognitive decline, with abnormal vital signs (e.g., fever, tachycardia) and lung examination findings. Diagnosis should be confirmed by chest radiography or ultrasonography." [15]
  * Chronic pulmonary obstructive disease exacerbation "An event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough, and/or sputum and beyond normal day-to-day variations, that is acute in onset and may warrant a change in regular medication in a patient with underlying COPD" [16]
  * Adult respiratory distress syndrome (Berlin definition)
  * Need for mechanical ventilation
  * Need for non-invasive mechanical ventilation
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | HFOT (High Flow With Tracheostomy Interface) | COT (Conventional Oxygen Therapy)
Number analyzed (Participants) | 24 | 25
Participants | 2 | 11

2. Secondary Outcome: Percentage of Patients Decannulated
Description: Number of patients who were decannulated prior to discharge.
Time Frame: 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow With Tracheostomy Interface | Conventional Oxygen Therapy
Number analyzed (Participants) | 24 | 25
Participants | 18 | 23

3. Secondary Outcome: Hospital Length of Stay
Description: Number of days from admission to hospital discharge.
Time Frame: 35 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Flow With Tracheostomy Interface | Conventional Oxygen Therapy
Number analyzed (Participants) | 24 | 25
days | 10.125 (6.2) | 10.88 (6.3)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 2 months after surgery.
Arm/Group | HFOT (High Flow With Tracheostomy Interface) | COT (Conventional Oxygen Therapy)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HFOT (High Flow With Tracheostomy Interface) (N=24) | COT (Conventional Oxygen Therapy) (N=25)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Elevated blood glucose levels requiring initiation or escalation of medical therapy, including initiation of a regular insulin sliding scale for glycemic control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT05362526/Prot_SAP_004.pdf